CLINICAL TRIAL: NCT04591899
Title: Clinical and Radiographic Outcomes of CAD/CAM Versus Conventionally Constructed Occlusal Splints in Patients With Temporomandibular Joint Disorders: A Randomized Clinical Trial
Brief Title: Clinical and Radiographic Outcomes of CAD/CAM vs Conventionally Constructed Occlusal Splints in Patients With Temporomandibular Joint Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maram Ahmed Taema, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23091988
Record Dates: First submitted 2020-10-04; First posted 2020-10-19 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD/CAM SS (Experimental)
  Interventions: Device: CAD/CAM splints
- Conventionally manufactured SS (Active Comparator)
  Interventions: Device: CAD/CAM splints

INTERVENTIONS:
Device: CAD/CAM splints — Each of the maxillary and mandibular cast will scanned alone and then both scanned together in the centric relation using FREEDOM HD scanner1.
  The CAD/ CAM splint will be designed using Exocad software; the design will be the same as the conventional one. The surveying will be done by the software and the under-cuts blocked.
  The splints will be printed using Dent2 3D printer and then cured using Dentcure. The CAD/CAM splints material will be hard resin from PhotoCentric 3D.

SUMMARY:
The aim of this study is to compare between digitally formed occlusal splints versus conventional occlusal splints in patients with TMDs regarding patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

- Patients' age ranging from 20 to 50 years.

TMDs according to the research diagnostic criteria (RDC) for TMD (RDC/TMD) and magnetic resonance imaging (MRI) for confirmation which include:

i. Painful TMJ audible and palpable click. ii. No functional mouth limitation. iii. TMJ tenderness. Fully dentate patients without any malocclusion and good oral hygiene. Co-operative patient that should show motivation to follow up.

Exclusion Criteria:

* Patients with systemic diseases which could affect TMJ, e.g., rheumatoid arthritis, osteoarthrosis, Myasthenia Gravis and fibromyalgia.
* Patients showing bony irregularities e.g. osteophyte as recorded by Magnetic resonance imaging.
* Patients taking analgesic, muscle relaxant, or anti-inflammatory drugs were excluded because such drugs could influence the results.
* Any condition that contra-indicates MRI such as patients with pacemakers in heart.
* Patients with removable dental prosthesis

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction, done by questionnaire having the visual analogue scale | 3 months
  The questionnaire includes the following aspects; headaches, face pain, jaw joint pain, jaw joint noises, mastication pain, neck pain, face tension, limitation of mouth opening, complaints during mastication, and teeth sensitivity at baseline 1 and 2 weeks after, then after 1,2 and 3 months. The questioner will be translated into Arabic language to be understood by the patients.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR